CLINICAL TRIAL: NCT04513301
Title: Efficacy and Safety of Sintilimab With or Without Radiotherapy in Chinse Patients With Recurrent or IV NSCLC (EGFR -, ALK -) After Failure of Platinum-based Chemotherapy: A Randomized, Controlled, Phase II Clinical Study
Brief Title: Efficacy and Safety of Sintilimab With or Without Radiotherapy in Patients With Recurrent or IV NSCLC (EGFR -, ALK -) After Failure of Platinum-based Chemotherapy: A Randomized,Open Labled, Phase II Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Cancer Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBI308 ZL001
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — sintilimab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab alone (Active Comparator): Sintilimab (200 mg q3w ×2cycle)
  Interventions: Drug: Sintilimab
- Sintilimab+Radiotherapy (Experimental): Sintilimab (200 mg q3w ×2cycle)+RT 50-60Gy/25-30f
  Interventions: Drug: Sintilimab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Sintilimab — Sintilimab (200 mg q3w ×2 cycle)
Radiation: Radiotherapy — RT 50-60Gy/25-30f
  Arms: Sintilimab+Radiotherapy

SUMMARY:
Lung cancer incidence and mortality have been increasing steeply in the past thirty years in the mainland of China. More than 80% of lung cancer is non-small cell lung cancer (NSCLC). More than 40% of NSCLC patients are found to be in stage IIIb or IV, which is not resectable. The 5-year survival rate for this group of patients is less than 5% in the SEER database. Currently, the NCCN guidelines recommend platinum-containing double-drug chemotherapy as the first- line standard of care for advanced NSCLC without driver gene mutations, and treatment options after failure of first-line chemotherapy are limited. Immune Checkpoint Inhibitors, ICIs provide new treatment options, and in addition, radiotherapy can also be used in selected patients with advanced NSCLC, especially in patients with oligo progression, where irradiation of the thoracic primary lesions can improve the patient's respiratory-related symptoms, reduce the tumor burden, improve the patient's quality of life, and prolong survival in some patients. Therefore, we propose that combination of immunotherapy and radiotherapy to the primary lesion for these patients, who are generally in good KPS status, may result in improved quality of life and prolonged survival. To date, there have been no clinical studies of immunotherapy combined with primary lesions radiation therapy in patients with advanced non-small cell lung cancer (driver gene-negative) after chemotherapy failure or recurrence, so we designed this prospective, randomized, controlled, investigator-initiated, phase II clinical study with the primary objective of evaluating the efficacy of combined immunotherapy and primary lesions radiation therapy in this patient population. This trial aims at investigating the feasibility and efficacy of this treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to the implementation of any test-related process.
2. Age ≥ 18 and ≤ 75.
3. Life expectancy exceeding 3 months.
4. Non-small cell lung cancer is confirmed histologically or cytologically (either as an initial diagnosis or a subsequent biopsy). However, the Sputum cytology results alone are unacceptable. Cytology results of tracheal brush test, tracheal flush fluid and needle aspiration puncture is acceptable.
5. The investigator confirms the presence of at least one measurable lesion according to the RECIST 1.1 criteria.
6. Patients with stage IV, or recurrent NSCLC with histologically or cytologically confirmed , according to the International Association for the Study of Lung Cancer and the Joint Committee on American Cancer Classification, 8th edition, TNM stage of lung cancer.
7. Patients confirmed by histological specimens not applicable to EGFR or ALK-targeted therapy (with documented evidence of no tumor EGFR sensitivity mutations and no ALK gene rearrangements).
8. Eastern Oncology Collaborative Group (ECOG) fitness status score of 0 or 1.
9. Have received at least one regimen of platinum-containing chemotherapy with tumor progression or inability to tolerate chemotherapy response in the most recent chemotherapy regimen.
10. Good hematopoiesis, defined as an absolute neutrophil count ≥1.5 × 109/L, platelet count≥100 × 109/L, blood Erythropoietin ≥ 90 g/L
11. Good liver function, defined as total bilirubin levels ≤ 1.5 times the upper limit of normal(ULN); in patients without hepatic metastases, glutinous rice cereal is used as a supplement.
12. Aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times ULN; for patients with documented liver metastases, AST and ALT levels ≤ 5 times ULN.
13. Good renal function, defined as serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance ≥ 60 ml/min (Cockcroft-Gault formula); urine protein less than 2+ on routine urinalysis, or 24-hour urine protein quantification < 1 g.
14. Good coagulation, defined as an International Standardised Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times ULN; if the subject is receiving anticoagulant therapy, provided that the PT is within the intended use range of the anticoagulant.
15. For female subjects of childbearing age, a negative urine or serum pregnancy test should be presented within 3 days prior to receiving the first study drug administration (Week 1, Day 1). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test will be requested.
16. If there is a risk of conception, both male and female patients need to use highly effective contraception (i.e., a method with a failure rate of less than 1% per year) and continue until at least 180 days after discontinuation of the trial treatment.

Exclusion Criteria:

1. Currently participating in an interventional clinical research treatment, or has received another investigational drug or used an investigational device within 4 weeks prior to the first administration of the drug.
2. Previously received an anti-PD-1, anti-PD-L1, or anti-PD-L2 drug or a drug that stimulates or synergistically inhibits another T-cell receptor (e.g., CTLA-4, OX-40, CD137).
3. Systemic systemic therapy with an anti-lung cancer indication with a proprietary Chinese medicine or immunomodulatory drug (including thymidine, interferon, interleukin, except for local use for pleural control) within 2 weeks prior to the first dose, or major surgery within 3 weeks prior to the first dose.
4. Previous experience of chest radiotherapy.
5. Palliative radiotherapy completed within 7 days prior to the first administration of the drug.
6. Presence of clinically active diverticulitis, abdominal abscesses, gastrointestinal obstruction.
7. Have received a transplant of a solid organ or blood system.
8. Presence of clinically uncontrollable pleural effusion/abdominal fluid.
9. Known severe allergic reaction (grade ≥3) to cedirizumab, or other immunotherapeutic agents.
10. Active autoimmune disease requiring systemic therapy (e.g., use of disease-modifying drugs, corticosteroids, or immunosuppressants) occurring within 2 years prior to the first dose of the drug. Alternative therapies (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency) are not considered systemic therapy.
11. Diagnosis of immunodeficiency or being on systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days prior to the first administration of the study; physiological doses of glucocorticoids (≤10 mg/day of prednisone or equivalent) are permitted.
12. Have not sufficiently recovered from toxicity and/or complications from any of the interventions prior to initiating treatment (i.e. ≤ grade 1 or at baseline, not including weakness or hair loss).
13. Diagnosis of other malignancies within 5 years prior to the first dose, with exceptions including radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radically resected carcinoma in situ.
14. Symptomatic central nerve metastases. Patients with asymptomatic brain metastases or stable symptoms after treatment of brain metastatic lesions may be enrolled in this study if all of the following criteria are met: measurable lesions outside the central nervous system; absence of midbrain, bridge, cerebellum, medulla oblongata or spinal cord metastases; maintenance of clinical stability for at least 2 weeks; and cessation of hormonal therapy 3 days prior to the first dose of study drug.
15. A history of non-infectious pneumonia requiring glucocorticoid therapy or current interstitial lung disease within 1 year prior to the first administration of the drug.
16. Active infections that require systemic treatment.
17. (a) The known existence of a mental illness or substance abuse condition that may affect compliance with the test requirements.
18. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1/2 antibody positive).
19. Note: Subjects with hepatitis B who meet the following criteria are also eligible for enrollment: HBV viral load must be <1000 copies/ml (200 IU/ml) prior to first dose and subjects should receive anti-HBV therapy to avoid viral reactivation throughout the duration of study chemotherapy drug therapy. Subjects with anti-HBc (+), HBsAg (-), anti-HB (-) and HBV viral load (-) do not need to receive prophylactic anti-HBV therapy but need to be monitored closely for viral reactivation.
20. Active HCV-infected subjects (HCV antibody-positive and HCV-RNA levels above the lower limit of detection).
21. Live vaccine within 30 days prior to first dose (Cycle 1, Day 1); NOTE: Injectable inactivated viral vaccine against seasonal influenza is allowed up to 30 days prior to first dose; however, live attenuated influenza vaccine for intranasal administration is not allowed.
22. Evidence of a medical history or illness that could interfere with the results of the trial, prevent the subject from participating throughout the study, abnormal values for treatment or laboratory tests, or other circumstances that, in the opinion of the investigator, make enrollment unsuitable.
23. Breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
objective reactive rate | 12-week
  12-week objective reactive rate (ORR)
adverse events | three year
  grade 3-5 adverse events acording CTCAE 5.0

SECONDARY OUTCOMES:
progression-free survival (PFS) in two groups | three year
  Progression-Free Survival PFS is defined as the time from randomization to progression or death. (Time to progression is a related, less-preferred end point wherein deaths without progression are censored observations rather than counted as events.)

CONTACTS AND LOCATIONS:
Overall Officials: Min Fan, Study Director — Fudan University
Locations (1):
- Fudan University shanghai cancer center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided